CLINICAL TRIAL: NCT04618419
Title: Internal Jugular Vein Sonogram Versus Electrical Cardiometry For Assessment Of Fluid Responsiveness In Adult Undergoing Coronary Artery Bypass Graft Surgery
Brief Title: IJV Sonogram VS Cardiometry in Fluid Responsiveness In CABG
Status: Completed | Type: Observational
Sponsor: Ahmed Abd El-Rahim Abd El-Hamid Hammad (Other)
Responsible Party: Sponsor-Investigator, Ahmed Abd El-Rahim Abd El-Hamid Hammad, Residentat department of anaesthesia and surgical intensive Care, Alexandria University
Organization: Alexandria University (Other)
Other Study IDs: IJVDI and fluid responsiveness
Record Dates: First submitted 2020-10-20; First posted 2020-11-06 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Ultrasound of IJV; Electrical Cardiometry
Keywords: CABG surgery; Internal jugular vein; stroke volume variation; TFC

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: internal jugular vein distensibility index — It is a prospective observational clinical study to correlate hemodynamic monitoring between Electrical Cardiometry and internal jugular vein distensibility index by sonogram

SUMMARY:
The primary aim of the study is to assess the reliability of predicting fluid responsiveness in adults undergoing coronary artery bypass graft surgery using sonogram of the internal jugular vein for assessment of vessel distensibility in relation to stroke volume variation (SVV) measaured by electrical cardiometry.

The secondary aim is to evaluate the ability of thoracic fluid content (TFC) measured by electrical cardiometry to be an additive value for the assessment of fluid responsiveness.

DETAILED DESCRIPTION:
Fluid management is one of the most important treatments for stabilizing hemodynamics in patients after cardiac surgery.Electrical Cardiometry is a method for the non-invasive determination of stroke volume (SV), cardiac output (CO), stroke volume variation (SVV) and other hemodynamic parameters in adults, children, and neonates based on measurement of thoracic electrical bioimpedance and has been validated against "gold standard" methods such as thermodilution method of deriving CO using a pulmonary artery catheter (PAC).

The IJV is, technically, much more easily accessible for sonographic visualization than the IVC, and measurement of the IJV does not require transesophageal echocardiography (TEE). Internal jugular vein distensibility index (IJVDI) has been studied in several studies but its reliability has not been well confirmed in patients during cardiac surgery.

This is a prospective observational study of adults undergoing coronary artery bypass graft surgery . The primary aim of the study is to assess the reliability of predicting fluid responsiveness in adults undergoing coronary artery bypass graft surgery using sonogram of the internal jugular vein for assessment of vessel distensibility in relation to stroke volume variation (SVV) measaured by electrical cardiometry.The secondary aim is to evaluate the ability of thoracic fluid content (TFC) measured by electrical cardiometry to be an additive value for the assessment of fluid responsiveness.

Volume responsiveness will be independently assessed by IJV sonogram and electrical cardiometry in following times

1. After induction of anesthesia.
2. After transfusing 6 ml / kg of hydroxyethyl starch (HES) 6% before sternotomy.
3. After closure of the sternum and transfusion of patient's blood.
4. Immediately before transferring the patient to ICU and stabilization of hemodynamic parameters by giving fluids needed to patient.
5. Immediately after transferring the patient to ICU and stabilization of hemodynamic parameters by giving fluids needed to patient.
6. After 2 hour of ICU admission.
7. Before weaning from mechanical ventilation Fluid responsiveness will be assessed by examining SVV with a threshold of the SVV = 12% allow discrimination between Responders and Non-responders

ELIGIBILITY:
Inclusion Criteria:

Adults (>18 years old) Able to provide advanced informed consent Planned for elective CABG surgery

Exclusion Criteria:

* Age < 18 years
* Severely reduced preoperative left ventricular ejection fraction < 40 %
* Significant cardiac arrhythmia.
* Significant valvular heart disease.
* Clinically evident pulmonary disease.
* Bilaterally inserted venous catheters (jugular or subclavian vein)
* History of radiotherapy or surgery of the neck region.
* Inability to obtain interpretable ultrasound images due to a difficult acoustic window.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Demographic data, hemodynamic parameters as heart rate (HR), and mean arterial blood pressure (MAP),CVP and urine output have been registered.
  Cardiac data derived from electrical cardiometry including: CO ,cardiac index( CI), stroke volume variation( SVV) and thoracic fluid content were also recorded.
  IJVDI by sonogram was assessed
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2019-12-25 (Actual); Study Completion 2020-01-05 (Actual)

PRIMARY OUTCOMES:
fluid responsiveness after fluid challenge | 24 hours from the start of surgery
  Correlation between SVV and IJVDI

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria university, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aronson S, Nisbet P, Bunke M. Fluid resuscitation practices in cardiac surgery patients in the USA: a survey of health care providers. Perioper Med (Lond). 2017 Oct 19;6:15. doi: 10.1186/s13741-017-0071-6. eCollection 2017. PMID 29075482
- [Background] Ma GG, Hao GW, Yang XM, Zhu DM, Liu L, Liu H, Tu GW, Luo Z. Internal jugular vein variability predicts fluid responsiveness in cardiac surgical patients with mechanical ventilation. Ann Intensive Care. 2018 Jan 16;8(1):6. doi: 10.1186/s13613-017-0347-5. PMID 29340792